CLINICAL TRIAL: NCT02544945
Title: Comparing 3-D Printed vs Standard Bolus for Breast Cancer Chest Wall Radiotherapy: A Feasibility Study Measuring Bolus Spatial Accuracy, Dosimetric Accuracy and Treatment Set-up Time
Brief Title: Comparing 3-D Printed vs Standard Bolus for Breast Cancer Chest Wall Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rob Rutledge (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Rob Rutledge, Staff Radiation Oncologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3DBolus
Record Dates: First submitted 2015-07-20; First posted 2015-09-09 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: Radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Bolus (Active Comparator): The radiotherapy treatment days when the standard bolus is used
  Interventions: Other: Standard bolus
- 3D printed bolus (Experimental): the radiotherapy treatment days when the 3D bolus is used
  Interventions: Other: 3D printed bolus

INTERVENTIONS:
Other: 3D printed bolus — Using the Cat Scan for treatment planning, a 3D plastic shell can be produced which is shaped exactly to the shape of the patient's chest wall. This shell will act as bolus - the substance that is placed on the skin during chest wall radiotherapy. The bolus allows the right dose of radiotherapy to get to the skin and the underlying chest wall.
  Arms: 3D printed bolus
Other: Standard bolus — A standard 5mm-thick piece of rubber is placed on the patient's chest wall
  Arms: Standard Bolus

SUMMARY:
This is a cohort study of 16 women undergoing post-mastectomy chest wall radiotherapy for breast cancer comparing two ways of modifying the radiation beam with bolus (a 5mm rubber substance placed on the skin to modify the radiation beam). The hypothesis is that 3D printed bolus will conform more closely to the chest wall than standard 5mm-thick standard bolus and thus lead to less chance of underdose or overdose of the skin. Each patient will receive the standard dose of radiotherapy, but half the treatments will use standard bolus and half the treatments will 3D printed bolus (ie each patient will act as is their own control). The primary outcome is the comparison of the amount of air under the bolus for each technique. Secondary outcome is the amount of time it takes to set up the patient for radiotherapy.

DETAILED DESCRIPTION:
1. Study Schema

   Intervention

   All subjects receive standard chest wall radiotherapy doses as follows:
   * Half the days no bolus is applied to the chest wall as per the standard of care
   * Half the days bolus is applied - alternating days between standard 5mm rubber bolus and the experimental 3D printed bolus.

   Primary and Secondary Outcomes Each subject acts as their own control comparing the standard rubber bolus with the 3D printed bolus in terms of
   * The volume of air-gap between the bolus and the chest wall skin
   * The time it takes the radiation therapists to set up the patient
   * The calculated versus measured dose on the skin

   Sample size 16 patients over 4 months
2. Background and Rationale

In Canada, 25,000 women are diagnosed with breast cancer each year. Approximately 20% of these women undergo mastectomy (removal of the entire breast) as part of their curative treatment program. Radiotherapy is administered to the chest wall (where the breast was) in women whose breast cancer has spread to the lymph nodes

or in other situations in which there is a high chance there might be microscopic amounts of cancer cells left over on the chest wall. A meta-analysis of 25 randomized trials involving 8505 lymph node positive women showed post-mastectomy radiotherapy improved 10-year chest wall control rates from 73% to 92.5%. The same overview showed 15-year overall survival increased by 5.4% (60.1 vs 54.7%) in those women undergoing radiotherapy compared to those who did not.

Applying radiotherapy evenly to the chest wall during a course of 16-25 daily radiation treatments is technically challenging because, without modification, the high-energy radiotherapy machines under-dose the superficial tissue (exactly where the cancer cells might reside). To compensate for this phenomenon, a flexible polymer (rubber) "bolus" layer 3-10 mm thick is placed on the skin of the chest wall on some or all days of a radiation course. All sorts of bolus are used internationally from rubber to candle wax slabs. This standard 'bolus', typically 40 cm wide by 40 cm long, is placed on the chest wall and kept in place with tape and straps for the 15 minutes it takes to set up and administer the radiotherapy each day the bolus is applied. Because the contour of each women's chest wall is different and often include 'peaks and valleys' in the tissue, there is inevitably some 'air gaps' between the skin and the bolus material. This air gap, as seen easily on set up imaging, varies from day to day because the radiation therapists can't reproduce the exact placement of bolus, and women undergoing treatment can't get back into the exact same position on the radiotherapy bed each day. The varying air gaps can affect how much radiotherapy is getting to the skin, and can produce potential under-dosing of the cancer cells or overdosing of the normal skin.

In the Department of Radiation Oncology in Halifax the investigators have developed an innovative solution to this problem of air gap by using a 3D printing technology to create bolus that will be tailored to the exact shape of a patient's chest wall. The investigators have approximately 3 years of experience in producing 3D printed bolus for radiotherapy applications, including rigorous assessment of spatial and dosimetric accuracy of the tissues underneath the bolus. Previous research focused on medical physics validation studies, producing a 'smart bolus' to tailor electron therapy treatments at multiple treatment sites. Through this work the investigators have demonstrated that printed bolus conforms precisely even to complex patient anatomy, based on realistic phantom studies (i.e., models of patients including challenging situations e.g., treating part of a foot or ear). The bolus is designed directly from the planning CT data the patient anatomy, which is required for each patient for usual treatment planning calculations. The 3D printed bolus is typically 5 mm thick for x-ray photon beam applications and consists of polylactic acid (PLA), which is derived from starches (corn, sugar tapioca), inert, and commonly used for e.g., drinking cups and surgical pins. The average density of 3D bolus is controllable during printing and thus the investigators are able to replicate the density of the standard rubber bolus material. The investigators have shown previously that the material is accurately accounted for by the treatment planning system as confirmed in another study.

A recent in-house study of 3D printed bolus of the thickness used for this study show the calculated and measured on the machine closely correlate.

In the proposed study, producing a 3D printed bolus for each patient's chest wall could produce multiple advantages over the current technique:

1. The 3D bolus may decrease the amount of air gap between the bolus and the skin. Air gap currently limits the accuracy and uniformity of delivered radiation therapy. The 3D printed bolus would be individualized for every patient and designed and fabricated with sub-millimeter precision;
2. The time required by multiple radiation therapists to prepare the bolus setup prior to CT imaging may be reduced, particularly for challenging anatomies, given that the 3D printed bolus is produced in an automated way from CT data afterwards (without the patient and therapists present).
3. The time to set up a patient on the treatment machine (linear accelerator) may be decreased if individualized bolus 'slips' into place (compared to status-quo where bolus positioning can be iterative, error-prone and time-consuming).
4. As each patient will have their own individualized bolus, issues of infection control (contamination of bacteria from reusing the standard bolus) will be mitigated.

3. Study Objectives

To test whether 3D printed bolus produces less air gap, is faster to apply, and produces a reliable buildup of radiotherapy compared with standard rubber bolus on women undergoing chest wall radiotherapy.

4. Study Methods

This is a single-centre study accruing breast cancer patients who have already agreed to undergo chest wall radiotherapy

Study Flow for an Individual Patient

1. Accrual of patient and completion of consent process
2. CT simulation and standard bolus production (done exactly as per current standard of care)
3. Production of 3D printed bolus using the Simulation CT scan
4. Choice of location and calculation of skin dose
5. Creation of an individualized patient treatment plan

   * Plan generated by dosimetrists - alternating bolus on and bolus off
   * Outline of which days will be standard bolus and 3D bolus
6. Delivery of Radiotherapy on No bolus days- as per standard of care
7. Delivery of Radiotherapy on Bolus days

   * Application of the Diodes to the Chest wall
   * Timing of Set up time
   * CBCT scan on machine for set up (allows for measurement of air gap afterwards)
8. Monitoring of patient while on and after treatment

   * Air gap calculation
   * Measured dose to the skin
   * Skin reaction

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing radiotherapy to the chest wall for the treatment of breast cancer with radical intent.

Exclusion Criteria:

* Patients in whom the Radiation Oncologist plans to either omit bolus for more than half of the treatments (rarely happens).
* Patients undergoing a non-standard chest-wall technique (eg. VMAT)
* Pregnant or plans to get pregnant during radiotherapy
* Inability to obtain informed consent or adhere to the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Air gap under bolus | Up to 3 month
  Air gap is defined as a) the greatest distance from the skin to the bolus measured perpendicular to the chest wall, and b) the maximal area of skin underlying the maximal air pocket

SECONDARY OUTCOMES:
Set up time | Up to 3 months
  Measured as the time it takes to lay the patient down on the radiotherapy table to the time it takes to finish placing the bolus.

CONTACTS AND LOCATIONS:
Overall Officials: Robert DH Rutledge, MD, Principal Investigator — Capital Health, Canada
Locations (1):
- NSHA-QEII Health Sciences Centre, Halifax, Nova Scotia, Canada